CLINICAL TRIAL: NCT02090972
Title: Evaluation of Past Medications in Older Patients With Fractures and Patients Hospitalized for a Non-surgical Reason.
Brief Title: The Impact of Opioids in Fractures - a Case Control Study
Acronym: FROP
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Collaborators: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Prof., Dr., Ruhr University of Bochum
Other Study IDs: FROP_BHL_Bochum
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Fractures
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with fracture: * fracture within the last 14 days
  * no other fractures within the last 6 month
  * patients >60 years
- Control Patients: * patients hospitalized for an internal reason
  * no other fractures within the last 6 month
  * patients >60 years

SUMMARY:
In this study, the risk of opioid medications on fractures in older adults is investigated. Patients from the surgical department with fractures and control patients from the internal department of the same hospital are inquired with a standardized questionaire about demographic and clinical risk factors for fractures. Osteoporotic fracture risk is assessed using quantitative ultrasound. An impact of recent opioid medications on fractures is hypothesised.

ELIGIBILITY:
Inclusion Criteria for both groups:

* age > 60 years
* written informed consent

Exclusion Criteria for both groups:

* malignant Disease within the last 12 month
* troubles with memory, dementia or Parkinsons disease
* other fractures within the last 6 month

Exclusion Criteria for the fracture group:

* alcoholised during the fall
* fracture older than 14 days

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalized patients in University Hospital, surgical and internal department
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Reported Opioid medication before hospital admission | interview: 20 min
  Standardized assessment of opioid medications taken before fracture or hospital admission to evaluate the impact of opioids in fractures.
  Exact doses, substances and intake habits are inquired.

SECONDARY OUTCOMES:
Bone density measures using Quantitative ultrasound (SAHARA) | 10 min
  Evaluation of fracture risk due to reduced bone density is performed using quantitative ultrasound.

CONTACTS AND LOCATIONS:
Locations (1):
- BG University Hospital Bergmannsheil, Ruhr University Bochum, Bochum, Germany